CLINICAL TRIAL: NCT01490710
Title: NAVADYN11 : Hemodynamic Impact of a New Ventilatory Support Mode With Diaphragmatic Synchronization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 11/6-H
Record Dates: First submitted 2011-12-07; First posted 2011-12-13 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Invasive Ventilatory Support
Keywords: NAVA; Hemodynamic; Cardiac Index; Children with admission weight > 5kg

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: collection of clinical and biological parameters — Investigation focal lies in hemodynamic monitoring during the last 10 minutes (Cardiac Index Assessment and clinico-biological parameters as: ventilatory and respiratory parameters, NIRS, GDS, Omega Score, heart rate, blood pressure, lactate, BNP, perfusion coefficient…)
Other: assign optimal ventilatory mode — End of study: At the end of the second session, clinician will assign optimal ventilatory mode regarding patient clinical response.

SUMMARY:
Despite spectacular advances since the 90s mechanical ventilation used in intensive care units are amply associated with cardio-respiratory complications: nosocomial pneumonia, lung parenchyma lesions induced by ventilation, hemodynamic instability and ultimately to a significant morbidity and mortality.

NAVA (Neurally Adjusted Assist Ventilation) ventilatory support, provides synchronous support, proportionate to patient's respiratory efforts. More "physiological", this mode would decline its efficacy on patient hemodynamic response. However, to date, no study has focused on hemodynamic impact of NAVA. This is precisely the purpose of NAVADYN11 study, which aims to assess NAVA efficacy on cardiac index in pediatric intensive care unit.

ELIGIBILITY:
Inclusion criteria:

* Servo-i with NAVA available at patient admission
* Sedation protocol compatible with NAVA functioning
* Parental consent

Non inclusion criteria:

* Digestive pathology incompatible with gastric tube.
* Deep sedation required defined by score ComfortB <11 (cranial traumatism…)
* Brain damage incompatible with spontaneous ventilation
* Duration of intubation too short for investigation

Exclusion criteria:

* Clinical worsening requiring treatment and/or management inconsistent with NAVADYN11 research (CPR, emergency surgery ...). However, the investigator is allowed to reiterate investigation when patient stabilized.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-11

PRIMARY OUTCOMES:
Assess the impact of NAVA ventilation on hemodynamic parameters
  Assess the impact of NAVA ventilation on hemodynamic parameters in children hospitalized in a Paediatric Intensive Care Unit. Endpoint evaluation consists in a non-invasive measurement of cardiac index by esophageal doppler.

SECONDARY OUTCOMES:
Omega score
  SaO2/SaO2-SvO2
Heart rate
Blood pressure
NIRS
Blood gas
Lactate
BNP
Perfusion score
Right cardiac work index
  if available

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas JORAM, Doctor, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Liet JM, Barriere F, Gaillard-Le Roux B, Bourgoin P, Legrand A, Joram N. Physiological effects of invasive ventilation with neurally adjusted ventilatory assist (NAVA) in a crossover study. BMC Pediatr. 2016 Nov 8;16(1):180. doi: 10.1186/s12887-016-0717-4. PMID 27821162